CLINICAL TRIAL: NCT00703599
Title: Phase I/II Study of Intravenous Administration of Activated Autologous Adipose-Derived Stromal Vascular Fraction in Patients With Type 1 Diabetes
Brief Title: Safety and Efficacy of Autologous Adipose-Derived Stem Cell Transplantation in Patients With Type 1 Diabetes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adistem Ltd (Industry)
Responsible Party: Bill Paspaliaris / Director, Adistem Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ad-003
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2008-07-01 (Estimated); Status verified 2008-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus; Adipose-derived stem cells; Adipose stromal vascular fraction; Autologous; Insulin-dependence
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): This is the only arm and that is the treatment group.
  Interventions: Procedure: Autologous Adipose-derived Stem cells

INTERVENTIONS:
Procedure: Autologous Adipose-derived Stem cells — Intravenous administration of autologous activated stromal vascular fraction derived from 100-120 ml lipoaspirate following mini-liposuction of abdominal adipose tissue.
  Other Names: Treatment Group

SUMMARY:
The purpose of this study is to determine whether intravenous administration of autologous adipose stem cells is safe and beneficial in patients with type 1 diabetes.

DETAILED DESCRIPTION:
Diabetes Mellitus is of large epidemic proportions worldwide. It is proliferating at such a fast rate that new novel drugs and other therapeutic approaches are required. The purpose of this Phase I/II study is to determine whether the intravenous administration of activated adipose-derived stromal vascular fraction as a single procedure is safe and efficacious in patients with Type 1 Diabetes Mellitus. Patients will be observed over 12 months following the procedure, with 2 weeks, 1 month and tri-monthly diagnostics and life style questionaires.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Type I diabetes for at least 2 years
* Insulin-dependent

Exclusion Criteria:

* Presence of acute diabetic complications in the acute stage as recent myocardial infarction, recent CVA or acute renal failure.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Lowering of insulin-dependence and anti-hyperglycemic medication dosages | At 2, 4, 12, 24, 36, and 48 weeks

SECONDARY OUTCOMES:
Lowering of glycosylated hemoglobin (HbA1C). | At 4, 12, 24, 36, and 48 weeks
Increased circulating C-Peptide levels | At 4, 12, 24, 36, and 48 weeks.
Increased general well-being of patients. | At 2, 4, 12, 24, 36, and 48 weeks.
No detrimental change seen in kidney function tests, liver function tests and other haematological parameters. | At 2, 4, 12, 24, 36, and 48 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Emeritta A Barrenechea, MD, Principal Investigator — Veterens Memorial Medical Centre, Philippines; Florencio Q Lucero, MD, Principal Investigator — University of Philippines, College of Medicine; Letitia Lucero-Palma, MD, Study Director — Far Eastern University-NRMF Hospital, Quezon City, Philippines; Bill Paspaliaris, PhD, Study Chair — Adistem Ltd, Hong Kong
Locations (2):
- Philippines (2):
  - Beverly Hills Medical Group, Makati City, Manila
  - Veterens Memorial Medical Centre, Quezon City, Manila

REFERENCES:
- [Background] Gimble JM, Katz AJ, Bunnell BA. Adipose-derived stem cells for regenerative medicine. Circ Res. 2007 May 11;100(9):1249-60. doi: 10.1161/01.RES.0000265074.83288.09. PMID 17495232